CLINICAL TRIAL: NCT07044492
Title: The Effectiveness of Empathy-Based Program on Empathy Level Among Nursing Assistants in Long-term Care Facility
Brief Title: Effect of Empathy-Based Program on Nursing Assistants in Long-term Care Facilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202203004
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Long-Term Care; Long-term Care Facility
Keywords: Virtual Reality; Randomized Controlled Trial; Nursing Assistants; Empathy-Based Program; Debriefing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors were masked to group assignments to reduce assessment bias. No other parties were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (VR) with debriefing Group (Experimental): Participants in this group will engage with immersive virtual reality (VR) with debriefing.
  Interventions: Behavioral: Virtual Reality (VR) with Debriefing
- Control Group (C) (No Intervention): Participants in this group will continue their usual care routine without additional exposure to virtual.

INTERVENTIONS:
Behavioral: Virtual Reality (VR) with Debriefing — Participants will receive a weekly 5-minute VR session featuring immersive experiences of residents' lives within the facility, followed by a 25-minute debriefing discussion in small groups of 5~6 participants. This will continue for three weeks.
  Arms: virtual reality (VR) with debriefing Group

SUMMARY:
This randomized controlled trial aims to explore the impact of an Empathy-Based Program on the level of empathy among nursing assistants in a long-term care facility. A total of 100 participants will be divided into two groups: a virtual reality (VR) with debriefing group, and a control group (C) receiving routine care. The intervention involves a weekly 5-minute VR session featuring immersive experiences of residents' lives within the facility, followed by a 25-minute debriefing discussion in small groups of 5~6 participants. This will continue for three weeks. The study will evaluate the effectiveness of the empathy program in enhancing nursing assistants' empathy levels, with data collection occurring at three time points: baseline, post-intervention, and one-month follow-up.

DETAILED DESCRIPTION:
This study aims to investigate whether an Empathy-Based Program can enhance the level of empathy among nursing assistants working in long-term care facilities. The trial will include 100 participants who will be randomly assigned to one of two groups: a virtual reality (VR) with debriefing group, and a control group (C) receiving routine care. The intervention consists of a 30-minute session once a week for three weeks, comprising a 5-minute virtual scenario video followed by a 25-minute small-group debriefing session with 5 to 6 participants.

The primary objective of the study is to assess the impact of the Empathy-Based Program on participants' empathy levels, empathic behaviors, and attitudes toward older adults. Data will be collected at multiple time points throughout the intervention, and statistical analyses will be conducted to determine the effectiveness of the empathy-based sessions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria:

  1. Possess a valid nursing assistant license
  2. Aged 20 years or older
  3. Have worked at a long-term care institution for more than 3 months
  4. Able to read and understand written Chinese

     Exclusion Criteria:
* Employed as a part-time nursing assistant

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Empathy level | Baseline (pre-intervention), end of intervention (week 3), and follow-up at one month post-intervention (week 7)
  This study will use the 20-item version of the Jefferson Scale of Empathy-Health Professions version (JSE-HP). The scale has 20 items scored on a 7-point Likert scale, ranging from 1 (minimum) to 7 (maximum), with a total score between 20 and 140. Higher scores indicate greater empathy level among nursing assistants.
Attitudes toward older people | Baseline (pre-intervention), end of intervention (week 3), and follow-up at one month post-intervention (week 7)
  This study will use the Chinese version of the Kogan's Attitudes toward Older People (KAOP) Scale, translated and validated by Yeh et al. (2009), to assess participants' attitudes toward older adults. The KAOP consists of 34 items, including 17 positively worded and 17 negatively worded statements. Each item is rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Negatively worded items are reverse-coded before computing the total score. The possible total score ranges from 34 to 238, with higher scores indicating more positive attitudes toward older people.
Empathic Behavior | Baseline (pre-intervention), end of intervention (week 3), and follow-up at one month post-intervention (week 7)
  This study will use a 12-item Empathic Behavior Scale developed by the researchers based on a review of relevant literature. The scale is designed to assess the frequency of empathic behaviors performed by nursing assistants in various caregiving scenarios. Each item presents a specific situation, and participants are asked to indicate how frequently they perform the described empathic behavior using a 7-point Likert scale, ranging from 1 (never able to perform) to 7 (always able to perform). Total scores range from 12 to 84, with higher scores indicating more frequent engagement in empathic behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: No